CLINICAL TRIAL: NCT04233242
Title: Genotype-Informed Versus Empiric Management of VirEmia (GIVE MOVE) in HIV-Infected Children and Adolescents on Antiretroviral Therapy: An Open-Label Randomised Clinical Trial
Brief Title: Genotype-Informed Versus Empiric Management of VirEmia
Acronym: GIVE MOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: University Hospital, Basel, Switzerland (Other); University of Basel (Other); SolidarMed, Partnerships for Health (Unknown); Seboche Mission Hospital (Unknown); Ifakara Health Institute (Other); Baylor College of Medicine Children's Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P001-20-1.4; REG-19-008 (Other Grant/Funding Number: Fondation Botnar); ID 229-2019 (Other: National Health Research Ethics Committee (Lesotho)); Req-2019-01275 (Other: Ethikkommission Nordwest- und Zentralschweiz (Switzerland)); 12-2020 (Other: Ifakara Health Institute Review Board (Tanzania)); NIMR/HQ/R.8a/Vol. IX/3222 (Other: National Institute for Medical Research (Tanzania)); TMDA0020/CTR/0003/03 (Other: Tanzania Medicines and Medical Devices Authority (Tanzania))
Record Dates: First submitted 2020-01-11; First posted 2020-01-18 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2023-04

CONDITIONS: HIV-1-infection
Keywords: HIV-1; acquired immunodeficiency syndrome; drug resistance; treatment failure; child; adolescent; Lesotho; Tanzania
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Multi-centre, open-label, parallel-group (1:1 allocation), superiority randomised clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The viral load ≥400 c/mL before enrolment triggers genotypic resistance testing (GRT), followed by GRT-informed patient management and counselling. Onward treatment is informed by the resistance profile determined through GRT, with a GRT Expert Committee issuing a treatment recommendation.
  Interventions: Other: Clinical management informed by HIV-1 genotypic resistance testing
- Control (No Intervention): Standard of care according to national guidelines and recommendations of the World Health Organization: The viral load ≥400 c/mL before enrolment is followed by 3 sessions of enhanced adherence counselling and a follow-up viral load test. Onward treatment is informed by viral load testing.

INTERVENTIONS:
Other: Clinical management informed by HIV-1 genotypic resistance testing — The study intervention will consist of the following components:
  1. Genotypic resistance testing (GRT);
  2. Review of GRT results by an expert committee providing a treatment recommendation;
  3. GRT-based decision on further therapy (switch or maintain current ART regimen; choice of regimen); and
  4. GRT-informed adherence support.
  Arms: Intervention

SUMMARY:
HIV infection can be effectively controlled with antiretroviral therapy (ART). However, children and adolescents living with HIV and receiving ART suffer high rates of treatment failure, predominantly caused by suboptimal adherence to therapy and/or viral drug resistance. While high-income countries routinely use genotypic resistance testing (GRT) to determine which drug combinations are likely to be effective, this diagnostic tool is relatively costly and labour-intensive and is not routinely available in most resource-limited settings.

GIVE MOVE is a multi-country (Lesotho, Tanzania) randomised clinical trial assessing if rapid GRT after detecting an unsuppressed viral load improves the clinical management and thus health outcomes for children and adolescents living with HIV. Children and adolescents with an unsuppressed viral load despite ART are enrolled and randomly allocated to a control or an intervention arm (50% of participants in each arm). The control arm receives care according to the current standard of care, consisting of three sessions of enhanced adherence counselling at monthly intervals, followed by a second viral load test. Onward treatment is informed by the outcome of this viral load test alongside empirical guidelines and clinical judgement. The intervention arm receives GRT and GRT-informed onward therapy. Participants in the intervention arm also receive three sessions of enhanced adherence counselling, which is informed by GRT results (i.e., if no drug resistance is detected, there is a high chance of suboptimal adherence to ART and this can be directly addressed).

This trial will assess if the rapid provision of GRT improves participants' health outcomes at 9 months after enrolment. A nested study will assess the cost and cost-effectiveness of GRT. Thus, this trial will provide evidence on whether the provision of GRT for children and adolescents with HIV should be prioritised in resource-limited settings.

DETAILED DESCRIPTION:
Background and rationale:

Children and adolescents living with HIV and receiving antiretroviral therapy (ART) suffer high rates of treatment failure, predominantly caused by suboptimal adherence to therapy and/or viral drug resistance. While high-income countries routinely use genotypic resistance testing (GRT) to select an optimal ART regimen, this diagnostic tool is not routinely available in many resource-limited settings.

Objective:

The GIVE MOVE trial assesses if rapid GRT after detection of an unsuppressed viral load in children and adolescents on ART improves health outcomes when compared to the current standard of care. Furthermore, a nested study will assess the cost-effectiveness of this intervention. Combined, these results will provide evidence on whether GRT should be prioritised for children and adolescents with HIV.

Study design:

GIVE MOVE is a multi-centre (several centres in 2 countries, Lesotho and Tanzania), parallel-group (1:1 allocation), open-label randomised clinical trial. Children and adolescents living with HIV with a viral load ≥400 c/mL are enrolled.

The control group is managed as per the current standard of care that follows the World Health Organization guidelines, i.e. three sessions of enhanced adherence counselling at monthly intervals, followed by a second viral load test and viral load-informed onward treatment.

In the intervention arm, participants receive GRT, a GRT-informed treatment recommendation by a GRT Expert Committee, and GRT-informed onward therapy, selecting the best locally available drugs according to the drug resistance profile.

The GIVE MOVE trial will compare clinical outcomes (mortality, morbidity, viral suppression; see the Primary Outcome section for the composite primary endpoint) at nine months. Assuming that 20% vs 35% reach the primary endpoint in the intervention vs control arm, and at a significance level of 5%, 276 participants (138 per arm) are required to reach 80% power.

In addition to clinical outcomes, the trial intends to assess the cost and cost-effectiveness of the intervention. The GIVE MOVE trial aims at informing future clinical guidelines on the management of paediatric HIV.

ELIGIBILITY:
Inclusion Criteria:

* In care in a study site
* Age ≥6 months and <19 years
* Latest HIV viral load result ≥400 c/mL
* On an unchanged ART regimen for ≥6 months
* Phlebotomy for latest viral load test <4 months before screening
* Consent given

Exclusion Criteria:

* Indication for treatment switch according to WHO guidelines at screening
* 1st enhanced adherence counselling (EAC) session initiated >2 weeks prior to screening
* Intention to transfer out of the study site (and not into a different study site) within 3 months after randomisation
* Already enrolled in another study if judged as non-compatible by the (Local) Principal Investigator
* Pregnant or breastfeeding at screening (no exclusion based on pregnancy or breastfeeding after enrolment)
* Acute illness requiring hospitalisation at screening (no exclusion based on hospitalisation after enrolment)
* Received a resistance test in the last 12 months

Ages: 6 Months to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 286 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-07-08 (Actual)

PRIMARY OUTCOMES:
Composite primary endpoint | At 9 months follow-up visit (window: 32-44 weeks)
  The composite primary endpoint is the occurrence of any one or more of the events i) death due to any cause during the follow-up period (36 weeks), ii) HIV- or ART-related hospital admission of ≥24 hours duration (possibly, probably or definitely related to HIV or ART, judged by the endpoint committee blinded to the study arm) during the follow-up period (36 weeks), iii) new clinical World Health Organization (WHO) stage IV event (excluding lymph node tuberculosis, stunting, oral or genital herpes simplex infection and oesophageal candidiasis; judged by the endpoint committee blinded to the study arm) during the follow-up period (36 weeks), and iv) no documentation of a suppressed viral load (<50 c/mL) at 9 months follow-up (window: 32-44 weeks). The primary endpoint will be assessed as an event ratio of participants reaching one or more of the composite endpoints.

SECONDARY OUTCOMES:
Proportion with death due to any cause | Within 36 weeks after baseline
  Proportion of participants confirmed dead during the follow-period among all participants enrolled.
Proportion with HIV- or ART-related hospital admission of ≥24 hours duration | Within 36 weeks after baseline
  Proportion of participants with HIV- or ART-related hospital admission of ≥24 hours duration (possibly, probably or definitely related to HIV or ART, judged by the endpoint committee) during the follow-up period among all participants enrolled.
Proportion with new clinical WHO stage IV event(s) (with some exclusions) | Within 36 weeks after baseline
  Proportion of participants with new clinical WHO stage IV event(s) (excluding lymph node tuberculosis, stunting, oral or genital herpes simplex infection and oesophageal candidiasis; judged by the endpoint committee) during the follow-up period among all participants enrolled.
Proportion without documentation of a suppressed viral load | At 9 months follow-up visit (window: 32-44 weeks)
  Proportion of participants without documentation of viral load <50 c/mL at 9 months among all participants enrolled.
Proportion lost to follow-up | At 9 months follow-up visit (window: 32-44 weeks)
  Proportion of participants with no documented clinic visit at 9 months among all participants enrolled.
Proportion with observed virologic failure | At 9 months follow-up visit (window: 32-44 weeks)
  Proportion of participants with a viral load ≥50 c/mL among all participants with a viral load result at 9 months.
Composite endpoint | 6 months (window: 20-28 weeks) after the decision on onward treatment
  This composite endpoint is the proportion of participants among all participants enrolled experiencing one or more of the events i) death due to any cause within 24 weeks of the decision on onward treatment, ii) HIV- or ART-related hospital admission of ≥24 hours duration (possibly, probably or definitely related to HIV or ART) within 24 weeks of the decision on onward treatment, iii) new clinical WHO stage IV event (excluding lymph node tuberculosis, stunting, oral or genital herpes simplex infection and oesophageal candidiasis) within 24 weeks of the decision on onward treatment, and iv) no documentation of a suppressed viral load (<50 c/mL) at 6 months (window: 20-28 weeks) after the decision on onward treatment. The decision on onward treatment is defined as the first visit after the follow-up viral load result or resistance test result becomes available in the control or intervention arm, respectively.

OTHER OUTCOMES:
Time to viral suppression | 3- (window: 10-14 weeks), 6- (window: 20-28 weeks), and 9-month (window: 32-44 weeks) study visit
  Time to achieving a viral load <50 c/mL; considering viral load testing done with samples from the 3-, 6- and 9-month study visit in both arms.
Proportion with drug regimen switches in the absence of major drug resistance mutations and/or non-switches in the presence of major drug resistance mutations | Baseline and 9-month (window: 32-44 weeks) study visit
  Proportion of participants with drug regimen switches in the absence of major drug resistance mutations and/or non-switches in the presence of major drug resistance mutations among all participants enrolled (as identified by Sanger sequencing, according to the Stanford HIV drug resistance database).
Proportion with new drug resistance mutations emerged within the study period | Change from baseline to 9-month (window: 32-44 weeks) study visit
  Proportion of participants with new drug resistance mutations emerged within the study period among all participants enrolled.

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus D Labhardt, MD, MIH, Study Chair — Swiss Tropical & Public Health Institute; Jennifer A Brown, PhD, Principal Investigator — Swiss Tropical & Public Health Institute; Thomas Klimkait, PhD, Study Director — University of Basel; Josephine Muhairwe, MD, MPH, Study Director — SolidarMed, Partnerships for Health; Buntshi P Kayembe, MD, Study Director — Baylor College of Medicine Children's Foundation Lesotho; Mosa M Hlasoa, MD, Study Director — Baylor College of Medicine Children's Foundation Lesotho; Isaac Ringera, MPH, RN, Study Director — SolidarMed, Partnerships for Health; Maja Weisser, MD, Study Director — Swiss Tropical & Public Health Institute; Ezekiel Luoga, MD, Study Director — Ifakara Health Institute; Tracy R Glass, PhD, Study Director — Swiss Tropical & Public Health Institute
Locations (10):
- Lesotho (6):
  - Seboche Mission Hospital, Seboche, Butha-Buthe
  - Baylor Clinic Leribe, Hlotse, Leribe District
  - Baylor Clinic Butha-Buthe, Butha-Buthe
  - Baylor Clinic Maseru, Maseru
  - Baylor Clinic Mohale's Hoek, Mohale's Hoek
  - Baylor Clinic Mokhotlong, Mokhotlong
- Tanzania (4):
  - One-Stop Clinic and Chronic Diseases Clinic (CDCI) at St Francis Referral Hospital, Ifakara, Morogoro
  - Mbagala Rangi Tatu Hospital, Dar es Salaam
  - Temeke Regional Referral Hospital, Dar es Salaam
  - Upendano Dispensary, Dar es Salaam

IPD SHARING:
Plan to Share IPD: Yes
Upon publication of the trial results, a subset of the key pseudo-anonymised individual participant data collected during the study, along with a data dictionary, will be made available through the data repository Zenodo. The full dataset will be made available upon request to the Division of Clinical Epidemiology at the University Hospital Basel and after signing a data confidentiality agreement.

REFERENCES:
- [Background] Brown JA, Ringera I, Luoga E, Cheleboi M, Kimera N, Muhairwe J, Kayembe BP, Molapo Hlasoa M, Kabundi L, Yav CWD, Mothobi B, Thahane L, Amstutz A, Bachmann N, Mollel GJ, Bresser M, Glass TR, Paris DH, Klimkait T, Weisser M, Labhardt ND. Genotype-Informed Versus Empiric Management Of VirEmia (GIVE MOVE): study protocol of an open-label randomised clinical trial in children and adolescents living with HIV in Lesotho and Tanzania. BMC Infect Dis. 2020 Oct 19;20(1):773. doi: 10.1186/s12879-020-05491-9. PMID 33076866
- [Result] Brown JA, Ringera IK, Luoga E, Bresser M, Mothobi B, Kabundi L, Ilunga M, Mokhele K, Isaac AB, Tsoaeli N, Mbaya T, Simba B, Mayogu K, Mabula E, Cheleboi M, Molatelle M, Kimera N, Mollel GJ, Sando D, Tschumi N, Amstutz A, Thahane L, Hlasoa MM, Kayembe BP, Muhairwe J, Klimkait T, Glass TR, Weisser M, Labhardt ND. Resistance-informed versus empirical management of viraemia in children and adolescents with HIV in Lesotho and Tanzania (GIVE MOVE trial): a multisite, open-label randomised controlled trial. Lancet Glob Health. 2024 Aug;12(8):e1312-e1322. doi: 10.1016/S2214-109X(24)00183-9. PMID 39030062
- See also: trial website — https://www.givemove.org/

DOCUMENTS (2):
  • Study Protocol (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/42/NCT04233242/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT04233242/SAP_001.pdf